CLINICAL TRIAL: NCT05878288
Title: Comprehensive and Deep Profiling in Cutaneous Squamous Cell Carcinomas to Unravel Treatment Efficacy in Immunotherapy Treated Patients
Brief Title: Deep sequencIng in Cutaneous Squamous CEll caRciNomas
Acronym: DISCERN
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Collaborators: University of Melbourne (Other); University of Adelaide (Other); Monash University (Other); Regeneron Pharmaceuticals (Industry); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HREC/88736/PMCC-2022-326880
Record Dates: First submitted 2023-04-17; First posted 2023-05-26 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Cutaneous Squamous Cell Carcinoma; Cutaneous Squamous Cell Carcinoma of the Head and Neck; Neoplasms; Non-melanoma Skin Cancer
Keywords: single-cell sequencing; molecular profiling; neoadjuvant; immunotherapy; cemiplimab
MeSH Terms: conditions — Neoplasms | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Cemiplimab (Other): Cemiplimab 350 mg intravenously every 3 weeks for up to 12 weeks (up to 4 doses), or until unacceptable toxicity, disease progression, or withdrawal of consent.
  Interventions: Drug: Cemiplimab

INTERVENTIONS:
Drug: Cemiplimab — Cemiplimab 50 mg/mL supplied as a sterile liquid in single-use glass vials.
  Other Names: Libtayo, REGN-2810, REGN2810, cemiplimab-rwlc

SUMMARY:
To comprehensively describe the molecular profile of the tumour ecosystem of cutaneous squamous cell carcinoma (CSCC) patients treated with neoadjuvant immunotherapy using single-cell sequencing and bulk genomic profiling.

DETAILED DESCRIPTION:
The purpose of this study is to comprehensively assess the molecular profile of the tumour ecosystem of CSCC patients who receive immunotherapy in the neoadjuvant curative setting, in order to identify molecular mechanisms facilitating treatment response and resistance and to identify molecular markers for disease monitoring. Patients who receive immunotherapy for the neoadjuvant management of CSCC will be invited to participate in this translational research study during their treatment journey to provide tumour tissue (fresh and formal-fixed paraffin-embedded, FFPE) and blood samples before and after exposure to immunotherapy.

This study has primarily a translational research objective with the clinical component conducted as a prospective, single-centre, single-arm, open label study.

ELIGIBILITY:
Inclusion Criteria:

1. Stage II to IV (M0) CSCC who are candidates for surgery, but who have an increased risk of recurrence and/or risk of disfigurement or loss of function. Patients with stage III or IV (M0) CSCC of the head/neck, extremity, or trunk are eligible, and patients with stage II CSCC (≥3 cm longest diameter in an aesthetically sensitive region).
2. At least one measurable lesion per RECIST 1.1.
3. Age ≥18 years.
4. Histologically confirmed diagnosis of invasive CSCC.
5. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
6. Anticipated life expectancy >12 weeks.
7. Adequate organ function defined as:

   i) Hepatic function:
   1. Total bilirubin ≤1.5× upper limit of normal (ULN).
   2. Patients with Gilbert's Disease and total bilirubin up to 3× ULN are eligible.
   3. Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) ≤3× ULN.
   4. Alkaline phosphatase (ALP) ≤2.5× ULN. ii) Renal function: Serum creatinine ≤2× ULN or estimated creatinine clearance >35 mL/min (according the method of Cockcroft and Gault). iii) Creatinine phosphokinase (CPK) (also known as CK [creatinine kinase]) elevation ≤ grade 2. iv) Bone marrow function:

   <!-- -->

   1. Haemoglobin ≥9.0 g/dL.
   2. Absolute neutrophil count (ANC) ≥1.5 x 109/L.
   3. Platelet count ≥75 x 109/L.

Exclusion Criteria:

1. Active solid malignancy or haematological malignancies including chronic lymphocytic leukaemia, (unless indolent or non-life-threatening) within the last 5 years. For clarity, exceptions include other non-melanoma skin cancer that has undergone potentially curative therapy, or in-situ cervical carcinoma or in-situ prostate cancer with non-detectable prostate specific antigen or any other tumour that has been treated, and the patient is deemed to be in complete remission for at least 2 years prior to enrolment.
2. Metastatic disease.
3. Steroid use >10mg prednisone per day within 14 days of study drug (except if physiologic replacement).
4. Active autoimmune disease requiring active systemic therapy within the last 5 years.
5. Interstitial lung disease or pneumonitis requiring systemic therapy in the last 5 years.
6. Active infection requiring therapy including human immunodeficiency virus (HIV)-1 or HIV-2 serum antibody, hepatitis B virus (HBV), or hepatitis C virus (HCV), or active tuberculosis.
7. Breast-feeding or positive serum pregnancy test consistent with pregnancy (excluding false positives defined as a failure of βHCG doubling in 48 hours) or inability to comply with recommended contraception.
8. Receipt of live vaccine (including attenuated) within 30 days of first study treatment.
9. Prior transplant recipient (corneal transplant patients are eligible).
10. Prior PD-L1/PD-1 inhibitor exposure for the same lesion as enrolment.
11. Squamous cell carcinoma of unknown primary (those with presumed clinical assessment of CSCC are eligible).
12. Any anticancer treatment other than radiation therapy (such as chemotherapy, targeted systemic therapy, imiquimod, photodynamic therapy), either investigational or standard of care, within 30 days of the initial administration of cemiplimab or planned to occur during the study period.
13. History of documented allergic reactions or acute hypersensitivity reaction attributed to antibody treatments.
14. Patients with allergy or hypersensitivity to cemiplimab or to any of the excipients must be excluded.
15. Institutionalised patients by order of judicial or administrative authority.
16. Not willing to comply with all study related procedures, particularly consent for collection of tumour and blood samples and imaging, at all protocol specified time points.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-05-26 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Rate of successful execution and generation of data from single-cell RNA sequencing and genomic profiling (including whole exome sequencing, RNA sequencing and immunohistochemistry) of CSCC from patients treated with immunotherapy | At 72 months
  Generation of analyzable data from single-cell RNA sequencing and genomic profiling

SECONDARY OUTCOMES:
To evaluate pathological response rates (cPR, mPR defined as <10% viable tumour, and other). | Estimated 48 months
To evaluate ORR using computed tomography (CT) scan imaging assessed by RECIST 1.1 | Estimated 48 months
To evaluate ORR using computed tomography (CT) scan imaging assessed by imRECIST | Estimated 48 months
To summarise immune-related adverse events (AE) > grade 2, AESI, AEs > grade 3 and SAEs, according to CTCAE v5.0. | At 72 months
To evaluate DFS rates. | Estimated 48 months
To evaluate OS rates. | Estimated 48 months

OTHER OUTCOMES:
To describe any changes in the extent of surgical plans with the use of neoadjuvant immunotherapy, comparing plans at baseline and following neoadjuvant therapy. | Estimated 48months
  This outcome will be descriptive.
Describe molecular mechanisms underlying resistance to immunotherapy in CSCC by comparing tumour and TME profiles from immunotherapy responders vs nonresponders defined using pathological response and CT imaging, to identify putative therapeutic targets. | 72 months
  The outcome will be descriptive.
Describe whether genomic changes identified in CSCC and TME are detectable in cfDNA and whole blood, and whether these correlate with treatment response. | 72 months
Describe molecular mechanisms underlying response to immunotherapy in CSCC by comparing tumour and TME profiles from immunotherapy responders vs nonresponders defined using pathological response and CT imaging, to identify putative predictive biomarkers. | 72 months

CONTACTS AND LOCATIONS:
Overall Officials: Annette M Lim, MBBS, FRACP, PhD, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (1):
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No